CLINICAL TRIAL: NCT01727934
Title: A Phase 2, Open-Label, Clinical Trial of Miravirsen Sodium in Null Responder to Pegylated-Interferon Alpha Plus Ribavirin Subjects With Chronic Hepatitis C (CHC) Virus Genotype 1 Infection
Brief Title: Miravirsen Study in Null Responder to Pegylated Interferon Alpha Plus Ribavirin Subjects With Chronic Hepatitis C
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPC3649-207
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C
Keywords: Antisense; miR-122 antagonist; host factor; Chronic hepatitis C; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — miravirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miravirsen sodium (Experimental): Miravirsen will be dosed as single subcutaneous injections. Subjects will receive 5 weekly doses at 7 mg/kg then 4 every other week doses at 5 mg/kg.
  Interventions: Drug: Miravirsen sodium

INTERVENTIONS:
Drug: Miravirsen sodium — Subcutaneous injection
  Other Names: SPC3649

SUMMARY:
The purpose of this open-label study is to assess the safety, antiviral activity, and pharmacokinetics of 9 subcutaneous injections of miravirsen monotherapy (5 weekly doses over 5 weeks, followed by a further 4 doses once every other week over 7 weeks) over a total of 12 weeks of treatment. The subjects enrolled in this study are chronically infected with HCV genotype 1 and are null responders to treatment with peg IFNα/RBV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hepatitis C
* HCV genotype 1
* BMI 18-38 kg/m2
* Null responder to pegylated interferon alpha and ribavirin

Exclusion Criteria:

* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Significant liver disease in addition to hepatitis C
* Decompensated liver disease medical history or current clinical features
* Histologic evidence of hepatic cirrhosis
* Concurrent clinically significant medical diagnosis (other than CHC)
* Concurrent social conditions (e.g. drugs of abuse, alcohol excess, poor living accommodation)
* Clinically significant illness within 30 days preceding entry into the study
* Participated in an investigational drug study within 30 days or 5 half-lives, whichever is longer, prior to the start of study medication
* History of clinically significant allergic drug reactions

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with sustained virological response 24 weeks after the end of therapy. | 36 weeks

SECONDARY OUTCOMES:
The proportion of subjects with a sustained virological response 12 and 48 weeks after the end of therapy. | 60 weeks
The proportion of subjects with undetectable HCV RNA levels at the end of treatment. | 12 weeks
Change in HCV RNA levels from baseline throughout the study. | 60 weeks
The proportion of subjects who experience virological failure throughout the study. | 60 weeks
Safety will be assessed by evaluation of adverse events, physical examinations, vital signs, 12-lead ECGs, and laboratory assessments (clinical chemistry, hematology, urinalysis). | 60 weeks

OTHER OUTCOMES:
Viral resistance analysis at baseline and throughout the study. | 60 weeks
  The miR-122 seed sites in HCV RNA from subjects at baseline and following viral breakthrough or relapse will be subjected to genotypic sequence analysis.
Plasma pharmacokinetics | 28 weeks
  Plasma PK for miravirsen levels will be determined for up to 2 hours post-dose on Day 1, up to 24 hours post-dose on Days 29 and 84, and pre-dose for all other treatment period visits. Additionally, plasma PK will be evaluated at all follow-up visits through Week 28.
Urine pharmacokinetics | Up to 24 hours post-dose on Day 29 and Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Maribel Rodriguez-Torres, MD, Principal Investigator — Fundacion de Investgacion de Diego
Locations (1):
- Fundacion de Investigation de Diego, San Juan, Puerto Rico